CLINICAL TRIAL: NCT00592527
Title: Evaluation of Insulin Detemir in Combination With OADs in Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy of Insulin Detemir in Combination With OADs in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1569
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir

SUMMARY:
This trial is conducted in Asia.

The aim of this trial is to evaluate the blood glucose achieved with insulin detemir as add-on to current oral antidiabetic drug (OAD) treatment in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months since diagnosis
* Insulin naive subjects
* OAD treatment for at least 4 months with max. two OAD treatments
* Body mass index below 30.0 kg/m2
* HbA1c between 7.0-11.0%

Exclusion Criteria:

* OAD treatment with three or more OADs
* Secondary diabetes
* Known hypoglycaemia unawareness or recurrent major hypoglycaemia as judged by the Investigator
* Uncontrolled hypertension
* Known or suspected allergy to trial product or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2004-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 20 weeks of treatment

SECONDARY OUTCOMES:
Fasting plasma glucose (FPG)
Within-subject variation
Change in body weight
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- India (4):
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Ahmedabad
  - Novo Nordisk Investigational Site, Chennai
  - Novo Nordisk Investigational Site, Nagpur

REFERENCES:
- [Result] Ramachandran A, Harish K, Sundaram A, Mayur P, Sunil GS, Srishyla MV. Improved Efficacy when Insulin Detemir is added to OADs in Indian Subjects with Type 2 Diabetes. Diabetes 2006; 55 (Suppl. 1): A469 (2028-PO)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com